CLINICAL TRIAL: NCT02598362
Title: Pharmacokinetics of Ciprofloxacin in Pediatric Patients With Emphasis on Renal Excretion
Brief Title: Pharmacokinetics of Ciprofloxacin in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-004638-24
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Urinary Tract Infection; Pyelonephritis
Keywords: ciprofloxacin; pharmacokinetics; excretion; clearance; infant; children; adolescent
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous (Other): Participants who are treated with ciprofloxacin intravenously, at discretion of the treating physician.
  Interventions: Drug: ciprofloxacin
- oral (Other): Participants who are treated with ciprofloxacin via the oral route, at discretion of the treating physician.
  Interventions: Drug: ciprofloxacin

INTERVENTIONS:
Drug: ciprofloxacin — Serum and urine concentrations after ciprofloxacin administration. pharmacokinetic testing after ciprofloxacin administration

SUMMARY:
Measuring serum and urine concentrations of ciprofloxacin after IV and oral administration in children aged 3 months - 17 years who are treated for urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

* age between 3 months and 17 years of age
* confirmed diagnosis of febrile urinary tract infection (a rectal body temperature of 38.5 °C.in combination with either significant leukocyturia or a positive urine nitrite test in a reliable urine sample.
* indication for treatment or uroprophylaxis with ciprofloxacin at discretion of the treating physician.

Exclusion Criteria:

* pregnancy
* impaired renal function as defined by 2x serum creatinine level for age and sex
* epilepsy
* myasthenia gravis
* long QT-syndrome
* glucose 6 phosphatase deficiency (G6PD)
* allergy to one of the substances of cipro
* concomitant use of corticosteroids
* for the oral group: co medication of antacidic drugs, ferrofumarate, calcium, magnesium or Zinc supplements.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Serum concentrations | 12 hours

SECONDARY OUTCOMES:
Urine concentrations | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Johan Vande Walle, MD PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - Ghent University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meesters K, Michelet R, Mauel R, Raes A, Van Bocxlaer J, Vande Walle J, Vermeulen A. Results of a Multicenter Population Pharmacokinetic Study of Ciprofloxacin in Children with Complicated Urinary Tract Infection. Antimicrob Agents Chemother. 2018 Aug 27;62(9):e00517-18. doi: 10.1128/AAC.00517-18. Print 2018 Sep. PMID 29987142